CLINICAL TRIAL: NCT02913326
Title: RE-SPECT CVT: a Randomised, Open-label, Exploratory Trial With Blinded Endpoint Adjudication (PROBE), Comparing Efficacy and Safety of Oral Dabigatran Etexilate Versus Oral Warfarin in Patients With Cerebral Venous and Dural Sinus Thrombosis Over a 24-week Period
Brief Title: A Clinical Trial Comparing Efficacy and Safety of Dabigatran Etexilate With Warfarin in Patients With Cerebral Venous and Dural Sinus Thrombosis (RE-SPECT CVT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.248; 2015-004412-38 (EudraCT Number)
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Dabigatran; Warfarin

ARMS (2):
- Dabigatran etexilate (Experimental)
  Interventions: Drug: Dabigatran etexilate
- Warfarin (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran etexilate
  Arms: Dabigatran etexilate
Drug: Warfarin
  Arms: Warfarin

SUMMARY:
This is a multi-center, prospective, international, randomized (1:1), open-label study with two parallel groups. This phase III study is planned to investigate the efficacy and safety of dabigatran etexilate versus dose-adjusted warfarin on a net clinical benefit endpoint of major bleeding (ISTH criteria) and new venous thrombotic event (VTE) (primary endpoint) with blinded endpoint adjudication.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent in accordance with International Conference on Harmonization (ICH) Good Clinical Practice (GCP) guidelines and local legislation and/or regulations
* Confirmed diagnosis of Cerebral Venous or dural sinus thrombosis (CVT), with or without intracranial haemorrhage
* Completion of anticoagulation therapy for 5-15 days which has been administered until randomisation; anticoagulation must include full-dose low molecular weight heparin or unfractionated heparin
* Eligibility for treatment with an oral anticoagulant
* Further inclusion criteria apply

Exclusion criteria:

* Cerebral Venous or dural sinus thrombosis (CVT) associated with central nervous system infection or due to head trauma
* Planned surgical treatment for CVT
* Conditions associated with increased risk of bleeding
* History of symptomatic non-traumatic intracranial haemorrhage with risk of recurrence according to Investigator judgment
* Treatment with an antithrombotic regimen for an indication other than CVT and requiring continuation of that treatment for the original diagnosis without change in the regimen
* Severe renal impairment
* Active liver disease
* Pregnancy, nursing or planning to become pregnant while in the trial
* Further exclusion criteria apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (36):
- France (2):
  - HOP Pellegrin, Bordeaux
  - HOP Lariboisière, Paris
- Germany (5):
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Universitätsklinikum Essen AöR, Essen
  - Asklepios Klinik Wandsbek, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Tübingen, Tübingen
- India (6):
  - Mazumdar Shaw Medical centre, Bangalore
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Caritas Hospital, Kottayam
  - Magnum Heart Institute, Nashik
  - All India Institute of Medical Sciences, New Delhi
  - Sahyadri Speciality Hospital, Pune
- Italy (6):
  - ASST di Cremona, Cremona
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Nuovo Ospedale Civile S. Agostino-Estense, Modena
  - A.O. San Camillo Forlanini, Roma
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
  - A. O. Ospedale Circolo Fond. Macchi, Varese
- Netherlands (2):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (4):
  - University Clinical Center, Gdansk, Gdansk
  - Copernicus Med.Company.Ltd,Hosp.Nicolaus, Gdansk, Gdansk
  - Independent Public Clin.Hospital No.4,Neurol.Dept,Lublin, Lublin
  - Psychiatry&Neurol.Instit.Interv.Stroke&Cerebrov.Treatm.Cntr, Warsaw
- Portugal (5):
  - Hospital Fernando Fonseca, EPE, Amadora
  - CHLO, EPE - Hospital Egas Moniz, Lisbon
  - CHULN, EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar São João,EPE, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E. - Hospital de São Sebastião, Santa Maria da Feira
- Russia (4):
  - Reg.State Budget Hlthcare,City Hosp#5,Neurology Dept,Barnaul, Barnaul
  - Interreg. Clinical & Diagnostic Center, Neurol. Dept., Kazan, Kazan'
  - St.Petersb,State Hlthcare Instit. Elisabeth Hosp,Neurol.dept, Saint Petersburg
  - Sverdlovsk Reg.Clin.Hosp.No.1, Yekaterinburg
- Spain (2):
  - Hospital Ramón y Cajal, Madrid
  - Hospital La Paz, Madrid

REFERENCES:
- [Derived] Ferro JM, Bendszus M, Jansen O, Coutinho JM, Dentali F, Kobayashi A, Aguiar de Sousa D, Neto LL, Miede C, Caria J, Huisman H, Diener HC; RE-SPECT CVT Study Group. Recanalization after cerebral venous thrombosis. A randomized controlled trial of the safety and efficacy of dabigatran etexilate versus dose-adjusted warfarin in patients with cerebral venous and dural sinus thrombosis. Int J Stroke. 2022 Feb;17(2):189-197. doi: 10.1177/17474930211006303. Epub 2021 Apr 4. PMID 33724104
- [Derived] Ferro JM, Coutinho JM, Jansen O, Bendszus M, Dentali F, Kobayashi A, van der Veen B, Miede C, Caria J, Huisman H, Diener HC; RE-SPECT CVT Study Group. Dural Arteriovenous Fistulae After Cerebral Venous Thrombosis. Stroke. 2020 Nov;51(11):3344-3347. doi: 10.1161/STROKEAHA.120.031235. Epub 2020 Sep 25. PMID 32972315
- [Derived] Ferro JM, Coutinho JM, Dentali F, Kobayashi A, Alasheev A, Canhao P, Karpov D, Nagel S, Posthuma L, Roriz JM, Caria J, Frassdorf M, Huisman H, Reilly P, Diener HC; RE-SPECT CVT Study Group. Safety and Efficacy of Dabigatran Etexilate vs Dose-Adjusted Warfarin in Patients With Cerebral Venous Thrombosis: A Randomized Clinical Trial. JAMA Neurol. 2019 Dec 1;76(12):1457-1465. doi: 10.1001/jamaneurol.2019.2764. PMID 31479105
- [Derived] Ferro JM, Dentali F, Coutinho JM, Kobayashi A, Caria J, Desch M, Fraessdorf M, Huisman H, Diener HC. Rationale, design, and protocol of a randomized controlled trial of the safety and efficacy of dabigatran etexilate versus dose-adjusted warfarin in patients with cerebral venous thrombosis. Int J Stroke. 2018 Oct;13(7):766-770. doi: 10.1177/1747493018778125. Epub 2018 May 18. PMID 29775170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomised, open-label, exploratory trial with blinded endpoint adjudication (PROBE [prospective, randomised, open-label, blinded endpoint] design), comparing efficacy and safety of oral dabigatran etexilate versus oral warfarin in patients with cerebral venous and dural sinus thrombosis over a 24-week period.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that they (all participants) met all inclusion/exclusion criteria. Participants were not to be randomised to trial treatment if any one of the specific entry criteria were not met.
Groups:
- Dabigatran Etexilate: Participants were orally treated with Dabigatran etexilate 150 milligram (mg) capsule twice daily for 24 weeks.
- Warfarin: Participants were orally treated with Warfarin 1 mg/3 mg/5 mg tablet, as needed to maintain a target international normalised ratio (INR) of 2.0 - 3.0, once daily for 24 weeks.
Period: Overall Study
Arm/Group | Dabigatran Etexilate | Warfarin
Started | 60 | 60
Completed | 59 | 58
Not Completed | 1 | 2
Not completed — Reason not listed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The set includes patients who received at least one dose of study medication and were analysed according to the treatment they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate | Warfarin | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.4 (14.06) | 46.0 (13.64) | 45.2 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 27 | 27 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 15
  Not Hispanic or Latino | 52 | 43 | 95
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 45 | 49 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite of Venous Thrombotic Event (VTE) or Major Bleeding Event (MBE) According to International Society on Thrombosis and Haemostasis (ISTH) Criteria in Full Observation Period.
Description: Composite of the percentage of participants with MBE according to ISTH criteria and VTE (recurring cerebral venous thrombosis (CVT); deep venous thrombosis (DVT) of any limb, pulmonary embolism (PE), splanchnic vein thrombosis) in full observation period. All components were adjudicated in a blinded manner.
  Major bleeds were defined according to the ISTH definition of a major bleed, as follows:
  * Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome and/or
  * Bleeding associated with a reduction in haemoglobin of at least 2 grams/deciLitre (1.24 millimole/Litre) within 24 h, or leading to transfusion of 2 or more units of blood or packed cells and/or
  * Fatal bleed
Time Frame: From first administration of trial medication until 6 days after last administration of trial medication, up to 25 weeks.
Population: Full analysis set (FAS): All patients randomised were analysed in the treatment group to which they were randomised regardless of whether they took study medication. This followed the intent-to-treat principle.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 60 | 60
Percentage of participants | 1.7 [0.0 to 8.9] | 3.3 [0.4 to 11.5]

2. Secondary Outcome: Percentage of Participants With Recurring Cerebral Venous and Dural Sinus Thrombosis; DVT of Any Limb, PE or Splanchnic Vein Thrombosis in Full Observation Period
Description: VTE criterions:
  * New neurological signs/symptoms or worsening of previous signs/symptoms with new CVT on neuroimaging.
  * DVT of any limb was documented by: Abnormal compression ultrasonography; An intraluminal filling defect on venography; At autopsy
  * Splanchnic vein thrombosis: The presence of endoluminal material/absence of flow in the extrahepatic portal veins/mesenteric veins as shown by duplex-Doppler ultrasound/contrast-enhanced CT scan/MRI.
  * PE was documented by: An intraluminal filling defect in segmental/more proximal branches on spiral CT scan; An intraluminal filling defect/an extension of an existing defect/a sudden cut-off of vessels>2.5 mm in diameter on the pulmonary angiogram; Perfusion defect of at least 75% of a segment with a local normal ventilation result on ventilation/perfusion lung scan; Inconclusive spiral CT, pulmonary angiography/lung scintigraphy with demonstration of DVT in the lower extremities by compression ultrasonography/venography; At autopsy.
Time Frame: as for outcome 1
Population: FAS,
  Magnetic resonance imaging (MRI), Computed tomography (CT)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 60 | 60
Percentage of participants
  Recurring CVT | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 6.0]
  DVT of any limb | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 6.0]
  PE | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 6.0]
  Splanchnic vein thrombosis | 0.0 [0.0 to 6.0] | 0.0 [0.0 to 6.0]

3. Secondary Outcome: Cerebral Venous Recanalisation as Measured by the Change in Number of Occluded Cerebral Veins and Sinuses at Week 24
Description: Cerebral venous recanalisation was assessed by imaging and was adjudicated. Occlusion of cerebral veins and sinuses was scored as: 1 = full occlusion; 0 = no occlusion/partial occlusion. This score was applied using the below conventions: Superior sagittal, straight, cavernous sinuses, left and right jugular veins each scored individually as either 0 or 1; Right lateral transverse and sigmoid sinus were scored together, Left lateral transverse and sigmoid sinus were scored together, Superior petrous sinus and inferior petrous sinus were scored together; Deep venous system, Superficial cortical veins, Cerebellar veins were scored as systems.
  For each patient a total score was calculated at baseline and at EOT and the recanalisation score was calculated as EOT - baseline total scores with conventions as 0 = no cerebral veins or sinuses fully occluded and 11 = all cerebral veins and sinuses fully occluded; the lower the score, the better.
Time Frame: Baseline and week 24
Population: FAS - Patients with missing/not analysable MRI scan at baseline or end of treatment (EOT) are excluded from the analysis
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 55 | 52
Units on scale | -0.8 (0.78) | -1.0 (0.92)

4. Secondary Outcome: Percentage of Participants With Major Bleeding According to ISTH Criteria in Full Observation Period
Description: Major bleeds were defined according to the ISTH definition of a major bleed, as follows:
  * Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome and/or
  * Bleeding associated with a reduction in haemoglobin of at least 2 grams/deciLitre (1.24 millimole/Litre) within 24 h, or leading to transfusion of 2 or more units of blood or packed cells and/or
  * Fatal bleed
Time Frame: as for outcome 1
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 60 | 60
Percentage of participants | 1.7 [0.0 to 8.9] | 3.3 [0.4 to 11.5]

5. Secondary Outcome: Composite Endpoint of Percentage of Participants With New Intracranial Haemorrhage or Worsening of the Haemorrhagic Component of a Previous Lesion After up to 24 Weeks
Description: Intracranial haemorrhage (ICH) comprised the subtypes of intracerebral bleeds, subdural bleeds, epidural bleeds and subarachnoid bleeds that were recorded.
Time Frame: From first administration of trial medication until end of treatment visit, up to 24 weeks.
Population: TS - Patients with missing/not analysable MRI scan at baseline or EOT are excluded from the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 56 | 53
Percentage of participants | 1.8 [0.0 to 9.6] | 3.8 [0.5 to 13.0]

6. Secondary Outcome: Percentage of Participants With Clinically Relevant Non-major Bleeding Events in Full Observation Period.
Description: A clinically relevant non-major bleeding event (CRNMBE) was a clinically overt bleed that did not meet the criteria for a major bleed but prompted a clinical response, in that it led to at least 1 of the following: A hospital admission (i.e. overnight stay in the hospital) for bleeding / A physician guided medical or surgical treatment for bleeding / A physician guided change, interruption or discontinuation of trial medication.
Time Frame: as for outcome 1
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 60 | 60
Percentage of participants | 0.0 [0.0 to 6.0] | 1.7 [0.0 to 8.9]

7. Secondary Outcome: Percentage of Participants With Major Bleeding According to ISTH Criteria or CRNMBEs After up to 24 Weeks
Description: Percentage of participants with major bleeding according to ISTH criteria or CRNMBEs after up to 24 weeks.
Time Frame: From first administration of trial medication until end of treatment visit, up to 24 weeks.
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 60 | 60
Percentage of participants | 1.7 [0.0 to 8.9] | 5.0 [1.0 to 13.9]

8. Secondary Outcome: Percentage of Participants With Any Bleeding Event After up to 24 Weeks
Description: Percentage of participants with any bleeding event after up to 24 weeks where any bleeding event is the sum of all major and non-major bleeding events.
Time Frame: From first administration of trial medication until end of treatment visit, up to 24 weeks.
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dabigatran Etexilate | Warfarin
Number analyzed (Participants) | 60 | 60
Percentage of participants | 20.0 [10.8 to 32.3] | 20.0 [10.8 to 32.3]

ADVERSE EVENTS:
Time Frame: From first administration of trial medication until 6 days after last administration of trial medication, up to 25 weeks.
Description: TS
Arm/Group | Dabigatran Etexilate | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 8/60 | 6/60
Other Adverse Events (participants affected / at risk) | 21/60 | 17/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (N=60) | Warfarin (N=60)
Pyelonephritis (Infections and infestations) | 0 | 1
Severe fever with thrombocytopenia syndrome (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Evans syndrome (Blood and lymphatic system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Intestinal haematoma (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
International normalised ratio fluctuation (Investigations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (N=60) | Warfarin (N=60)
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Headache (Nervous system disorders) | 10 | 8
Depression (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT02913326/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02913326/SAP_001.pdf